CLINICAL TRIAL: NCT00102804
Title: A Phase 3, Double-Blind, Placebo-Controlled Study of Maintenance Pemetrexed Plus Best Supportive Care Versus Best Supportive Care Immediately Following Induction Treatment for Advanced Non-Small Cell Lung Cancer
Brief Title: Pemetrexed and Best Supportive Care Versus Placebo and Best Supportive Care in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5122; H3E-MC-JMEN (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pemetrexed and Best Supportive Care (Experimental)
  Interventions: Drug: Pemetrexed; Other: Best Supportive Care
- Placebo and Best Supportive Care (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: Pemetrexed — 500 milligrams per square meter (mg/m^2), intravenous (IV) administration, every (q) 21 days, until disease progression
  Other Names: LY231514; Alimta
  Arms: Pemetrexed and Best Supportive Care
Drug: Placebo — IV administration, q 21 days
  Arms: Placebo and Best Supportive Care
Other: Best Supportive Care — Treatment without a specific antineoplastic regimen, given with the intent to maximize quality of life, as judged by the treating physician.

SUMMARY:
This study is a randomized Phase 3, double-blind study of maintenance pemetrexed plus best supportive care versus placebo plus best supportive care in NSCLC. Participants must have received 1 of 6 induction regimens for 4 cycles and did not have progressive disease prior to randomization (enrollment) into this trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC Stage IIIB (with pleural effusion and/or positive supraclavicular lymph nodes) or Stage IV prior to induction therapy.
* Participants must have had 1 of the following induction therapies for treatment for Stage IIIB (with pleural effusion and/or positive supraclavicular lymph nodes) or IV NSCLC: Gemcitabine plus carboplatin, paclitaxel plus carboplatin, or docetaxel plus carboplatin, gemcitabine plus cisplatin, paclitaxel plus cisplatin or docetaxel plus cisplatin.
* Participants must have received only 1 chemotherapeutic doublet lasting precisely 4 cycles.
* Induction regimens must be based on 21-day cycles.
* Documented evidence of a tumor response of complete response (CR), partial response (PR), or stable disease (SD). Tumor assessment must occur between Cycle 4 (Day 1) of induction therapy and the date of randomization. This response does not have to be confirmed in order for the participant to be randomized. Positron emission tomography (PET) scans and ultrasounds may not be used for lesion measurements for response determination.

Exclusion Criteria:

* With the exception of those chemotherapies listed as inclusion criterion, participants will not be included if they have received prior systemic anticancer therapy (including adjuvant early-stage treatment for NSCLC) or any systemic treatment for any other cancer.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that would compromise the participant's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2005-03; Primary Completion 2007-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (73):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portsmouth, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshfield, Wisconsin
- Australia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bankstown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coffs Harbour, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Macquarie, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nambour, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Townsville, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashford, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ijuí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Bulgaria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varna
- China (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dalian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb, Croatia
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava-Poruba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chania
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mosdós
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szombathely
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banglagore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., P.O Ernakulam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Italy (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Livorno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Messina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ede
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zutphen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwolle
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Spain (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcorcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcoy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mataró
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murcia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Cruz de Tenerife
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei, Taiwan
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir

REFERENCES:
- [Derived] Belani CP, Brodowicz T, Ciuleanu TE, Krzakowski M, Yang SH, Franke F, Cucevic B, Madhavan J, Santoro A, Ramlau R, Liepa AM, Visseren-Grul C, Peterson P, John WJ, Zielinski CC. Quality of life in patients with advanced non-small-cell lung cancer given maintenance treatment with pemetrexed versus placebo (H3E-MC-JMEN): results from a randomised, double-blind, phase 3 study. Lancet Oncol. 2012 Mar;13(3):292-9. doi: 10.1016/S1470-2045(11)70339-4. Epub 2012 Feb 14. PMID 22336221
- [Derived] Gridelli C, Brodowicz T, Langer CJ, Peterson P, Islam M, Guba SC, Moore P, Visseren-Grul CM, Scagliotti G. Pemetrexed therapy in elderly patients with good performance status: analysis of two phase III trials of patients with nonsquamous non-small-cell lung cancer. Clin Lung Cancer. 2012 Sep;13(5):340-6. doi: 10.1016/j.cllc.2011.12.002. Epub 2012 Jan 23. PMID 22266043
- [Derived] Ciuleanu T, Brodowicz T, Zielinski C, Kim JH, Krzakowski M, Laack E, Wu YL, Bover I, Begbie S, Tzekova V, Cucevic B, Pereira JR, Yang SH, Madhavan J, Sugarman KP, Peterson P, John WJ, Krejcy K, Belani CP. Maintenance pemetrexed plus best supportive care versus placebo plus best supportive care for non-small-cell lung cancer: a randomised, double-blind, phase 3 study. Lancet. 2009 Oct 24;374(9699):1432-40. doi: 10.1016/S0140-6736(09)61497-5. Epub 2009 Sep 18. PMID 19767093
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who signed the informed consent form (ICF) and completed the randomized process are presented in the participant flow by the treatment arm to which they were randomized. Participants who did not sign the ICF or complete the randomization process were removed from the database and excluded from all analyses.
Groups:
- Pemetrexed and BSC: Pemetrexed: 500 milligrams per square meter (mg/m^2), intravenous (IV) administration, every (q) 21 days, until disease progression.
  Best Supportive Care (BSC): Treatment without a specific antineoplastic regimen, given with the intent to maximize quality of life, as judged by the treating physician.
- Placebo and BSC: Placebo: IV administration, q 21 days, until disease progression.
  BSC: Treatment without a specific antineoplastic regimen, given with the intent to maximize quality of life, as judged by the treating physician.
Period: Overall Study
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Started | 441 | 222
Received at Least 1 Dose of Study Drug | 434 | 222 (Four participants randomized to placebo received pemetrexed.)
Completed | 0 | 0
Not Completed | 441 | 222
Not completed — Progressive Disease (PD) | 307 | 196
Not completed — Withdrawal by Subject | 46 | 7
Not completed — Adverse Event | 37 | 3
Not completed — Physician Decision | 24 | 6
Not completed — Death | 5 | 6
Not completed — Enrollment Criteria Not Met | 6 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Satisfactory Response | 2 | 0
Not completed — Sponsor Decision | 1 | 0
Not completed — Alive, Receiving Treatment | 7 | 2

BASELINE CHARACTERISTICS:
Population: Participants who signed the ICF and completed the randomized process are reported according to the treatment arm to which they were randomized.
Groups:
- Pemetrexed and BSC: Pemetrexed: 500 mg/m^2, IV administration, q 21 days, until disease progression.
  BSC: Treatment without a specific antineoplastic regimen, given with the intent to maximize quality of life, as judged by the treating physician.
- Placebo and BSC: Placebo: IV administration, q 21 days.
  BSC: Treatment without a specific antineoplastic regimen, given with the intent to maximize quality of life, as judged by the treating physician.
- Total: Total of all reporting groups
Arm/Group | Pemetrexed and BSC | Placebo and BSC | Total
Number analyzed (Participants) | 441 | 222 | 663
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.6 [54.3 to 67.5] | 60.4 [53.8 to 67.0] | 60.6 [54.1 to 67.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 61 | 180
  Male | 322 | 161 | 483
Race/Ethnicity, Customized [Number; unit: participants]
  Aboriginal | 0 | 1 | 1
  African | 6 | 0 | 6
  Caucasian | 279 | 149 | 428
  East Asian | 104 | 50 | 154
  Hispanic | 13 | 6 | 19
  West Asian | 39 | 16 | 55
Region of Enrollment [Number; unit: participants]
  United States | 20 | 12 | 32
  Taiwan | 5 | 4 | 9
  Greece | 18 | 9 | 27
  Spain | 30 | 19 | 49
  Turkey | 7 | 4 | 11
  Austria | 2 | 2 | 4
  Italy | 18 | 16 | 34
  India | 39 | 16 | 55
  Hungary | 8 | 6 | 14
  Czech Republic | 5 | 2 | 7
  Poland | 25 | 11 | 36
  Brazil | 24 | 10 | 34
  Croatia | 10 | 3 | 13
  Romania | 51 | 26 | 77
  Australia | 19 | 8 | 27
  Bulgaria | 11 | 8 | 19
  Netherlands | 10 | 4 | 14
  Germany | 40 | 16 | 56
  China | 62 | 37 | 99
  Korea, Republic of | 37 | 9 | 46

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Time
Description: PFS time was the elapsed time from the date of randomization to the first date of objective progression of disease or death from any cause. PFS was censored at the date of the participant's last tumor assessment for participants who were not known to have died or to have PD as of the data-inclusion cut-off date for analysis. PD, defined using Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0), was at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Randomization to measured PD or death from any cause (up to 41 months)
Population: Participants who signed the ICF and completed the randomized process are reported according to the treatment arm to which they were randomized. Participants censored: N = 123, 36 participants in the pemetrexed and placebo treatment arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Number analyzed (Participants) | 441 | 222
months | 4.27 [4.07 to 4.73] | 2.60 [1.68 to 2.83]

2. Secondary Outcome: Overall Survival (OS) Time
Description: OS time was the elapsed time from the date of randomization to the date of death from any cause. OS was censored at the last date of contact for participants who were not known to have died as of the data-inclusion cut-off date for analysis.
Time Frame: Randomization to date of death from any cause (up to 41 months)
Population: Participants who signed the ICF and completed the randomized process are reported according to the treatment arm to which they were randomized. Participants censored: N = 138, 48 participants in the pemetrexed and placebo treatment arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Number analyzed (Participants) | 441 | 222
months | 13.37 [11.93 to 15.87] | 10.58 [8.74 to 12.02]

3. Secondary Outcome: Time to Objective Progressive Disease (TPD)
Description: TPD was the elapsed time from the date of randomization to the first date of objective PD. TPD was censored at the date of the participant's last tumor assessment for participants who were not known to have PD as of the data-inclusion cut-off date for analysis or who died without objective PD. PD, defined using RECIST v1.0, was at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Randomization to measured PD (up to 41 months)
Population: Participants who signed the ICF and completed the randomized process are reported according to the treatment arm to which they were randomized. Participants censored: N = 145, 40 participants in the pemetrexed and placebo treatment arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Number analyzed (Participants) | 441 | 222
months | 4.27 [4.11 to 4.73] | 2.60 [1.68 to 2.83]

4. Secondary Outcome: Time to Worsening of Symptoms (TWS)
Description: TWS was the elapsed time from the date of randomization to the first date of worsening [defined as a 15-millimeter (mm) increase from baseline based on a 100-mm scale] of each symptom and summary item in the Lung Cancer Symptom Scale (LCSS). The participant-reported LCSS was a 9-item questionnaire. Six items were symptom-specific measures for lung cancer (loss of appetite, fatigue, cough, dyspnea, hemoptysis, and pain), and 3 summation items described total symptomatic distress, interference with activity level, and global quality of life. Participant (pt) responses to each item were measured using visual analogue scales (VAS) from 0 (for best outcome) to 100 (for worst outcome). TWS was censored at the date of the last LCSS assessment for pts who were not known to have LCSS worsening.
Time Frame: Randomization to worsening of each LCSS item (up to 39 months)
Population: Pts who signed ICF and completed randomization, according to treatment randomized. Pts censored: Loss of appetite 236,140; fatigue 237,130; cough 274,146; dyspnea 271,143, hemoptysis 404,198; pain 271,135; symptom distress 247,141; interference with activity level 267,141, global quality of life 262,137 pts in pemetrexed, placebo arm, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Number analyzed (Participants) | 441 | 222
months
  Loss of appetite | 3.78 [2.86 to 4.44] | 4.40 [2.96 to 15.61]
  Fatigue | 3.06 [2.63 to 5.29] | 3.09 [2.43 to 3.98]
  Cough | 6.05 [4.21 to 7.82] | 4.67 [3.06 to 15.61]
  Dyspnea | 5.36 [4.21 to 10.87] | 4.40 [2.83 to 15.61]
  Hemoptysis | NA [NA to NA] — Median (95% confidence interval) TWS for hemoptysis was not calculated due to the high level of censoring. | NA [NA to NA] — Median (95% confidence interval) TWS for hemoptysis was not calculated due to the high level of censoring.
  Pain | 6.11 [4.57 to 9.56] | 4.63 [3.32 to 5.98]
  Symptomatic distress | 4.21 [3.58 to 5.55] | 3.78 [2.99 to 18.53]
  Interference with activity level | 6.51 [4.34 to 8.18] | 3.98 [2.83 to 15.61]
  Global quality of life | 5.75 [4.37 to 8.41] | 3.71 [2.99 to 5.49]

5. Secondary Outcome: Percentage of Participants With a Complete Response (CR) or Partial Response (PR) (Objective Tumor Response Rate)
Description: Response was defined using RECIST v1.0 criteria. CR was defined as the disappearance of all target lesions. PR was defined either A) at least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LDs or B) complete disappearance of target lesions, with persistence (but not worsening) of 1 or more nontarget lesions. In either case, no new lesions may have appeared. The percentage of participants with CR or PR=(Number of participants with CR or PR)/(Number of participants assessed)*100.
Time Frame: Baseline to measured PD (up to 41 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Number analyzed (Participants) | 441 | 222
percentage of participants | 6.8 [5 to 10] | 1.8 [0 to 5]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Clinically significant events were defined as serious adverse events (SAEs) and other non-serious AEs regardless of causality. A summary of serious and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion (up to 41 Months)
Population: Participants who signed the ICF, completed the randomized process and received at least 1 dose of study drug are reported according to the treatment to which they were received.
Measure: Number; unit: participants
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Number analyzed (Participants) | 438 | 218
participants
  SAEs | 83 | 31
  Other Non-Serious AEs | 386 | 178

7. Secondary Outcome: Maximum Improvement Over Baseline in Individual Symptom Scores and Quality of Life Using the LCSS
Description: The participant-reported LCSS was a 9-item questionnaire. Six items were symptom-specific measures for lung cancer (loss of appetite, fatigue, cough, dyspnea, hemoptysis, and pain), and 3 summation items described total symptomatic distress, interference with activity level, and global quality of life. Participant responses to each item were measured using VAS from 0 (for best outcome) to 100 (for worst outcome). The average symptom burden index (ASBI) was the mean of the 6 symptom-specific items. The LCSS total score was the mean of the 9 items.
Time Frame: Baseline through 30 days post discontinuation of study treatment (up to 39 Months)
Population: Participants who signed the ICF, completed the randomization process, had LCSS data at baseline and at least once postdose are reported according to the treatment arm to which they were randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Number analyzed (Participants) | 403 | 197
units on a scale
  Loss of appetite (n=403, 197) | 7.3 (25.90) | 10.6 (25.25)
  Fatigue (n=403, 197) | 10.2 (27.10) | 10.4 (23.92)
  Cough (n=402, 197) | 7.6 (20.09) | 6.7 (23.81)
  Dyspnea (n=400, 196) | 7.6 (22.50) | 5.4 (20.44)
  Pain (n=401, 197) | 5.4 (20.96) | 4.3 (21.93)
  Hemoptysis (n=402, 196) | 1.5 (9.41) | 2.1 (9.23)
  Symptom distress (n=401, 196) | 6.5 (21.13) | 8.2 (22.5)
  Interference with activity level (n=400, 197) | 10.8 (27.08) | 9.3 (25.50)
  Global quality of life (n=401, 195) | 10.7 (24.94) | 10.5 (22.98)
  ASBI (n=392, 195) | 3.7 (12.34) | 3.8 (13.24)
  Total LCSS (n=388, 193) | 4.07 (12.76) | 4.04 (13.03)

ADVERSE EVENTS:
Description: Participants are reported under the treatment to which they received.
Arm/Group | Pemetrexed and BSC | Placebo and BSC
Serious Adverse Events (participants affected / at risk) | 83/438 | 31/218
Other Adverse Events (participants affected / at risk) | 386/438 | 178/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pemetrexed and BSC (N=438) | Placebo and BSC (N=218)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 3 (3)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 1/321 (1) | 0/158 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena caval occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pemetrexed and BSC (N=438) | Placebo and BSC (N=218)
Anaemia (Blood and lymphatic system disorders) | 65 (97) | 12 (15)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 25 (64) | 5 (8)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 21 (66) | 5 (5)
Neutrophilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (29) | 2 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (4) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Conjunctivitis (Eye disorders) | 20 (24) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Eye swelling (Eye disorders) | 2 (2) | 0 (0)
Eyelid oedema (Eye disorders) | 3 (3) | 0 (0)
Keratoconjunctivitis sicca (Eye disorders) | 4 (4) | 0 (0)
Lacrimation increased (Eye disorders) | 20 (21) | 0 (0)
Ocular surface disease (Eye disorders) | 3 (5) | 1 (2)
Photophobia (Eye disorders) | 2 (2) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 8 (10) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 18 (18) | 8 (8)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 3 (11)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 59 (85) | 17 (22)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 52 (88) | 15 (17)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 13 (18) | 6 (21)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 1 (2)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (7) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (5) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 102 (209) | 22 (24)
Odynophagia (Gastrointestinal disorders) | 4 (5) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 2 (4) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 19 (22) | 1 (1)
Tongue black hairy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 56 (88) | 9 (12)
Asthenia (General disorders) | 48 (74) | 10 (11)
Axillary pain (General disorders) | 2 (2) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 3 (14) | 0 (0)
Chest pain (General disorders) | 44 (67) | 16 (17)
Chills (General disorders) | 7 (9) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 6 (7) | 2 (2)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 145 (227) | 49 (63)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 7 (9) | 0 (0)
Influenza like illness (General disorders) | 10 (17) | 3 (4)
Injection site reaction (General disorders) | 4 (4) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 4 (4) | 0 (0)
Malaise (General disorders) | 2 (4) | 0 (0)
Mucosal inflammation (General disorders) | 12 (19) | 2 (2)
Obstruction (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 12 (16) | 1 (1)
Oedema peripheral (General disorders) | 27 (34) | 2 (3)
Pain (General disorders) | 24 (28) | 13 (13)
Peripheral coldness (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 56 (78) | 25 (33)
Swelling (General disorders) | 1 (1) | 0 (0)
Visceral oedema (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 6 (8) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 15 (17) | 2 (2)
Candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Cystitis (Infections and infestations) | 2 (3) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 3 (3)
Influenza (Infections and infestations) | 10 (12) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 14 (17) | 3 (3)
Oral candidiasis (Infections and infestations) | 4 (4) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Pyothorax (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (20) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (7) | 4 (4)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase decreased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 60 (87) | 9 (11)
Aspartate aminotransferase increased (Investigations) | 52 (63) | 8 (10)
Blood albumin decreased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase (Investigations) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 12 (16) | 4 (4)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine decreased (Investigations) | 3 (10) | 1 (1)
Blood creatinine increased (Investigations) | 21 (30) | 4 (4)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (3) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 9 (15) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (2) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 18 (28) | 2 (2)
Forced expiratory volume decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 6 (7) | 5 (5)
Glomerular filtration rate (Investigations) | 1 (3) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 5 (10) | 0 (0)
Granulocyte count decreased (Investigations) | 1 (1) | 0 (0)
Granulocyte count increased (Investigations) | 0 (0) | 1 (2)
Haemoglobin (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 19 (30) | 2 (2)
Neutrophil count decreased (Investigations) | 11 (16) | 1 (1)
Neutrophil count increased (Investigations) | 3 (4) | 0 (0)
Platelet count (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 5 (5) | 2 (2)
Platelet count increased (Investigations) | 1 (1) | 2 (3)
Red blood cell count decreased (Investigations) | 2 (5) | 1 (1)
Red blood cell microcytes present (Investigations) | 0 (0) | 1 (1)
Renal function test abnormal (Investigations) | 1 (3) | 0 (0)
Sensory level (Investigations) | 1 (1) | 0 (0)
Total bile acids increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Troponin t (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 17 (20) | 3 (3)
Weight increased (Investigations) | 5 (5) | 1 (1)
White blood cell count decreased (Investigations) | 4 (5) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 2 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alcohol intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 124 (238) | 40 (43)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (20) | 6 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (48) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 10 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (17) | 5 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (14) | 9 (11)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 4 (4)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 5 (6) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cognitive disorder (Nervous system disorders) | 2 (2) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 3 (3) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 34 (39) | 7 (7)
Dysaesthesia (Nervous system disorders) | 1 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 10 (14) | 1 (1)
Dysphasia (Nervous system disorders) | 2 (2) | 0 (0)
Formication (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 51 (62) | 19 (26)
Hemicephalalgia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 5 (6) | 3 (3)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 4 (4) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 10 (11) | 2 (2)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 27 (29) | 11 (12)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 22 (22) | 6 (6)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (2) | 0 (0)
Stupor (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0)
Depressed mood (Psychiatric disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 9 (9) | 1 (1)
Insomnia (Psychiatric disorders) | 28 (31) | 8 (8)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (8) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 5 (5) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 1/321 (1) | 0/158 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1/321 (1) | 0/158 (0)
Testicular pain (Reproductive system and breast disorders) | 1/321 (1) | 0/158 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/117 (2) | 0/60 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 95 (118) | 47 (50)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 98 (118) | 43 (45)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 10 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (23) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (6) | 4 (4)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 (15) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (22) | 7 (8)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 62 (81) | 14 (16)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Pneumatic compression therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 8 (10) | 5 (7)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 11 (11) | 4 (4)
Hypotension (Vascular disorders) | 6 (6) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Superior vena caval occlusion (Vascular disorders) | 3 (3) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Four participants (pts) assigned to placebo received pemetrexed; pts analyzed for efficacy as randomized. Three treated pts did not sign ICF, 1 treated pt signed ICF but did not complete entire randomization process; pts excluded from all analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days